CLINICAL TRIAL: NCT00451165
Title: Outcome Study of Bowel, Urinary and Sexual Function After Laparoscopic Colorectal Surgery, Using Questionnaire and Function Tests
Brief Title: Bowel, Urinary and Sexual Function After Laparoscopic Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: Kyoto University (Other)
Organization: Kyoto University Hospital (Other)
Other Study IDs: E-282
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2009-01

CONDITIONS: Surgery, Laparoscopic; Sexual Dysfunction, Physiological; Colorectal Surgery
Keywords: Laparoscopic; Colon; Rectal; Surgery; Urinary function; Sexual function; Bowel function; Male
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- colon
  Interventions: Procedure: laparoscopic colorectal surgery
- rectum
  Interventions: Procedure: laparoscopic colorectal surgery

INTERVENTIONS:
Procedure: laparoscopic colorectal surgery — laparoscopic colorectal surgery
  Other Names: endoscopic surgery

SUMMARY:
Research Populations: Male patients scheduled for laparoscopic colorectal surgery

Study Method: Questionnaire and function tests

Hypothesis: A laparoscopic nerve-sparing operation is not inferior to reported open surgery in preserving urinary and sexual function.

DETAILED DESCRIPTION:
There have been some reports that laparoscopically assisted rectal resection is associated with a higher rate of male sexual dysfunction compared with the open approach. But these reports are studied retrospectively.

We examine the frequency of bowel, urinary and sexual dysfunction prospectively in patients who received laparoscopic colorectal surgery.

We examine before operation, 7 days after, 3 months after, 6 months after and 12 months after operation, by questionnaires (International Index of Erectile Function (IIEF) 、Short Form-8 (SF8)、International Consultation on Incontinence Questionnaire-Short Form(ICIQ-SF)、International Prostate Symptom Score(IPSS)、Gastro-Intestinal Functional Outcome(GIFO)) and function tests (uroflowmetry and US).

ELIGIBILITY:
Inclusion Criteria:

* Male
* Laparoscopic right colon resection/laparoscopic rectal surgery
* 20-80 years old
* ECOG performance status (PS) 0-2

Exclusion Criteria:

* Emergent operation
* Previous proctectomy
* Severe urinary dysfunction

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients who will receive laparoscopic colorectal surgery
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2007-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiharu Sakai, Professor, Study Chair — Kyoto University Hospital
Locations (1):
- Kyoto University Hospital, Kyoto, Kyoto, Japan